CLINICAL TRIAL: NCT01888016
Title: Effectiveness of Fascial Manipulation in Early Rehabilitation Treatment of Rotator's Cuff Surgery Patients. A Randomized Trial.
Brief Title: Effectiveness of Fascial Manipulation in Rotator's Cuff Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manifa
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-08

CONDITIONS: Cuff Rotator Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fascial manipulation (Experimental)
  Interventions: Other: fascial manipulation; Other: standard physiotherapies treatment
- standard treatment (Active Comparator)
  Interventions: Other: standard physiotherapies treatment

INTERVENTIONS:
Other: fascial manipulation — • 3 manual intervention on deep fascial tissues, according to fascial manipulation technique, providing a specific motor and manual assessment, and a deep manual intervention over specific fascial alteration.
  Arms: fascial manipulation
Other: standard physiotherapies treatment — 10 standard treatments in 2 weeks
  * Deltoid and infraspinatus muscles electrotherapy
  * Chair for passive continue mobilization at allowed range of motion (ROM). ½ h per day
  * Scar massage
  * Upper limb, cervical spine and scapula massages
  * Passive and assisted/active shoulder mobilization exercises
  * Scapula micro-mobilizations
  * Gleno-humeral decoaptation
  * Elbow, wrist and hand active mobilization
  * Proprioceptive exercise with and without the aid of the mirror

SUMMARY:
The purpose is to evaluate the effectiveness of fascial manipulation treatment in terms to reduce pain and improve physical functionality after rotator's cuff surgery. The technique involves deep friction manipulation of fascia's specific spots. Distant from surgical site.

DETAILED DESCRIPTION:
To evaluate the effectiveness of fascial manipulation treatment associated with standard physiotherapies treatment in rotator's cuff surgery patients, we'll randomize about 60 patients for arm's of study. Both arm's will receive 10 standard physiotherapies treatments in 2 weeks while the experimental arm will receive 3 manual intervention on deep fascial tissues, according to fascial manipulation technique, providing a specific motor and manual assessment, and a deep manual intervention over specific fascial alteration.

To evaluate the effectiveness of fascial manipulation treatment we'll use 2 type of outcome measure and we will compare the result of both arms of study.

ELIGIBILITY:
Inclusion Criteria:

* Rotator's cuff surgery patients that have been operated within the past 4/5 weeks
* Age between 18 to 65 years old

Exclusion Criteria:

* Patients with traumatic shoulder's injury that involved bone's fractures.
* Severe underlying pathologies like rheumatic, neurological and cardio pathologies that affect the correct shoulder treatment
* Patients on anticoagulant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS)mean | Change from baseline in pain at the end of the rehabilitation cycle (two weeks)
  we'll compare the baseline data (the first evaluation), with data at the end of the treatment, and with follow up (30 days from surgery)

SECONDARY OUTCOMES:
Constant Murley score | Change from baseline in range of motion at the end of the rehabilitation cycle (two weeks)
  Constant Murley score for range of motion and shoulder function assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, MD, Study Chair — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy